CLINICAL TRIAL: NCT02611466
Title: A Phase 2a, Randomized, Double-blind, Placebo- and Naproxen Controlled, Parallel-group Study to Assess the Analgesic Efficacy of ASP7962 in Patients With Pain Due to Osteoarthritis of the Knee
Brief Title: A Study to Assess the Analgesic Efficacy of ASP7962 in Patients With Pain Due to Osteoarthritis of the Knee
Acronym: OAK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7962-CL-0022; 2014-004996-22 (EudraCT Number)
Record Dates: First submitted 2015-11-19; First posted 2015-11-20 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Osteoarthritis of the Knee; Chronic Lower Back Pain
Keywords: Osteoarthritis; ASP7962
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ASP7962 (Experimental): Participants receive 100 mg of ASP7962 orally twice daily for 4 weeks.
  Interventions: Drug: ASP7962
- Naproxen (Active Comparator): Participants receive 500 mg of naproxen orally twice daily for 4 weeks.
  Interventions: Drug: Naproxen
- Placebo (Placebo Comparator): Participants receive placebo orally twice daily for a period of 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP7962 — Participants receive ASP7962 100 mg orally twice daily, in the morning and evening with or without food (approximately 12 hours).
  Arms: ASP7962
Drug: Naproxen — Participants receive naproxen 500 mg orally twice daily, in the morning and evening with or without food (approximately 12 hours).
  Arms: Naproxen
Drug: Placebo — Participants receive matching placebo orally twice daily, in the morning and evening with or without food (approximately 12 hours).
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the analgesic efficacy of ASP7962 relative to placebo.

This study will also evaluate the efficacy of ASP7962 relative to placebo on pain on walking, function and stiffness; the time course of efficacy of ASP7962 relative to placebo; the improvement in overall patient status of ASP7962 relative to placebo as well as the safety and tolerability of ASP7962 relative to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a primary diagnosis of OA of the index knee with symptoms for at least 6 months prior to screening and patient meets American College of Rheumatology clinical classification criteria for OA of the knee, defined by the following:

  * Knee pain and at least 3 of the following 6:

    1. Age > 50 years
    2. Morning stiffness < 30 minutes
    3. Crepitus on active motion
    4. Bony tenderness
    5. Bony enlargement
    6. No palpable warmth of synovium
* Patient has a radiographic image of the index knee (according to the minimum quality criteria for radiographic image as set by the central radiology reader) showing evidence of OA with a Kellgren-Lawrence grade ≥2 at screening (based on central reading).
* Patient has moderate to severe index knee pain (pain due to OA of the knee at least 5 days per week for the last 3 months prior to screening, as determined by patient's medical history).
* Patient is ambulatory and the index knee must not contain any orthopedic and/or prosthetic device.
* WOMAC pain subscale score (with a 48-hour recall period) in the index knee ≥ 4 at baseline (visit 2 predose, mean of all questions on pain subscale).
* WOMAC physical function subscale score ≥ 4 at baseline (visit 2 predose, mean of all questions on physical function subscale with a 48-hour recall period).
* Patient is willing to discontinue all current pain medications during the baseline and treatment periods (until day 57) (except for allowed rescue medications). Low dose aspirin for cardioprophylaxis is allowed.
* Patient is compliant with daily pain recording. Compliance with diary completion will be defined as daily average pain ratings on at least 5 days of the baseline period, of which at least 3 days are in the last 4 days prior to visit 2.
* Male patient and their female spouse/partners who are of childbearing potential must be using a barrier method and 1 form of highly effective birth control starting at screening and continuing throughout the study period and for 90 days after the final study drug administration.
* Male patient must not donate sperm starting at screening and throughout the study period and for 90 days after the final study drug administration.
* Female patient must either:

  * Be of non-childbearing potential: post-menopausal (defined as at least 1 year without any menses) prior to screening, or documented surgically sterile
  * Or, if of childbearing potential: agree not to try to become pregnant during the study and for 28 days after the final study drug administration, and have a negative pregnancy test at screening and at baseline (visit 2 predose), and if heterosexually active, agree to consistently use a barrier method and 1 form of highly effective birth control starting at screening and continuing throughout the study period and for 28 days after the final study drug administration.
* Female patient must agree not to breastfeed starting at screening and continuing throughout the study period and for 28 days after the final study drug administration.
* Female patient must not donate ova starting at screening and continuing throughout the study period and for 28 days after the final study drug administration.
* Patient agrees not to participate in another investigational study from screening through the follow-up period (until day 57).

Exclusion Criteria:

Medical History / Clinical Status:

* Patient has a history of suicide attempt or suicidal behavior. Suicidal ideation within the last 12 months (a response of "yes" to questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale [C-SSRS]), or who are at significant risk to commit suicide, as judged by the investigator at screening and at the time of randomization.
* Patient has current or prior psychosis, major depressive disorder or other clinically significant psychiatric disorder.
* Patient has a current or prior clinically significant neurologic disease, including but not limited to peripheral neuropathy, stroke, cognitive impairment and seizure. Childhood febrile seizures are not exclusionary.
* Patient has any clinically significant uncontrolled musculoskeletal disorder (with the exception of OA), cardiovascular, gastrointestinal, endocrinologic (diabetes mellitus is allowed if controlled [glycated hemoglobin (HbA1c) ≤ 8.0%] and no peripheral neuropathy), hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, dermatologic, renal and/or other major disease.
* Patient has an active malignancy or a history of malignancy (except for treated nonmelanoma skin cancer) within the past 5 years.
* Patient has a history of inflammatory arthritis, (including rheumatoid arthritis or a history of RPOA, osteonecrosis or avascular necrosis of bone and/or joints), or has other diagnoses that may increase the risk of RPOA (e.g., pre-existing atrophic OA, subchondral insufficiency fracture), or severe knee malalignment or any other joint-related condition that makes the patient unsuitable for study participation (e.g., joint pain that is disproportionately severe, or which has atypical features for OA pain, should trigger further medical evaluation to rule out subchondral insufficiency fracture).
* Patient has findings suggestive of RPOA or increased risk for RPOA on screening radiographs of either index or non-index joints (based on central reading).
* Patient has a history of shoulder surgery, clinically significant trauma or current symptoms, including pain or impaired range of motion at shoulder joint.
* Patient has a coagulopathy, is receiving anticoagulants or has been diagnosed with thrombocytopenia or a functional platelet disorder.
* Patient has a history of paracetamol intolerance, or existence of medical condition or use of concomitant medication for which paracetamol is contraindicated.
* Patient has any contraindication to naproxen including but not limited to:

  * Known hypersensitivity to tramadol (a patient with intolerance or hypersensitivity is allowed, if the patient accepts to limit rescue medication toparacetamol).
  * Asthma, rhinitis, nasal polyps, urticarial or allergic-type reactions after taking aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs).
  * Anticipated coronary artery bypass graft surgery during the study.
  * Active or history of peptic ulceration.
  * Active or history of gastrointestinal bleeding (with the exception of hemorrhoids) or perforation.
* Patient has any contraindication to tramadol including but not limited to

  * Known hypersensitivity to tramadol.
  * Patient has used a monoamine oxidase inhibitor within 2 weeks prior to screening or during the screening or baseline periods.
* Patient has a body mass index (BMI) > 39 kg/m2.

Cardiovascular:

* Patient has a clinically significant abnormality on 12-lead electrocardiogram (ECG) at screening or baseline (visit 2 predose).
* Patient has any of the following:

  * Lifetime history of ischemic or hemorrhagic stroke, cardiac arrest, torsade de pointes, clinically significant structural heart disease or a personal or family history of long QT syndrome.
  * Within 12 months prior to visit 2: acute coronary syndrome (e.g., myocardial infarction, unstable angina [ischemic heart disease is allowed]); transient ischemic attack; coronary or peripheral revascularization procedure; clinically significant cardiac arrhythmias (including atrial fibrillation or flutter), heart block (first degree heart block is allowed provided PR interval is not greater than 240 msec) or other clinically significant cardiovascular disorder.
  * Current heart failure (New York Heart Association [NYHA] class III and IV).
* Patient has a resting pulse rate < 50 or > 100 beats per minute (bpm); systolic blood pressure (SBP) > 160 mm Hg; diastolic blood pressure (DBP) > 90 mm Hg at screening or baseline (visit 2 predose). These assessments may be repeated once, after a reasonable time period at the investigator's discretion. If the repeat measurement is meeting the above criteria, the patient will be excluded.
* Patient has a history of unexplained syncopal events or has symptomatic orthostatic hypotension at screening or baseline (visit 2 predose), defined as postural related symptoms and at least one of the following: standing SBP ≥ 20 mm Hg lower than supine SBP, standing DBP ≥ 10 mm Hg lower than supine DBP.

Clinical Chemistry / Hematology:

* Patient has (according to the investigator) clinically significant abnormalities in clinical chemistry, hematology or urinalysis at screening. These assessments may be repeated once, after a reasonable time period at the investigator's discretion (but within the screening period).
* Patient has any liver tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], total bilirubin [TBL]) > 1.5 times the upper limit of normal [ULN] at screening. These assessments may be repeated once, after a reasonable time period at the investigator's discretion (but within the screening period).
* Patient has an estimated glomerular filtration rate of ≤ 60 mL/min/1.73m2 (Modification of Diet in Renal Disease [MDRD] calculation) at screening.
* Patient has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis A virus antibodies (immunoglobulin M) (anti-HAV [IgM]), hepatitis C virus antibodies (anti-HCV), or antibodies to human immunodeficiency virus type 1(HIV-1) and/or type 2 (HIV-2) at screening.

Prior Medication / Medical Intervention:

* Patient has received any investigational drug within 28 days (or 5 half-lives of the investigational drug, whichever is longer) before screening or is scheduled to receive an investigational drug other than blinded study treatments during the course of this study.
* Patient has previously received antibodies to NGF within 3 months prior to screening.
* Patient has had any major surgery or orthopedic surgery within 3 months before screening or has plans for surgical intervention during the study.
* Patient who is not a suitable candidate for joint replacement surgery and who is unable to stop chronic NSAID use.
* Patient has received intra-articular corticosteroid or intra-articular local anesthetics within 3 months prior to screening, intra-articular hyaluronic acid within 6 months prior to screening or any of these therapies during the screening or baseline periods.
* Patient has received systemic corticosteroids within the past 30 days before screening or during the screening or baseline periods (topical, nasal and inhaled corticosteroids are permitted.)
* Patient has received any medications or nonmedication therapy with efficacy in reducing pain of OA of the knee, including over-the-counter (OTC) products (with the exception of ice packs, rest, and paracetamol) during the baseline period.
* Patient has started or stopped physiotherapy, acupuncture or transcutaneous electrical nerve stimulation related to treatment of the index knee within 4 weeks prior to screening or during the screening or baseline periods. Stable regimens of these therapies introduced more than 4 weeks prior to screening will be allowed if the regimen is to continue unchanged during the study.
* Patient has used opioids for more than 4 days during the week preceding screening or during the screening period; or has received any opioids during the baseline period.
* Patient has used dipeptidyl peptidase 4 (DPP-4) inhibitors within 12 months prior to visit 2.
* Patient has regularly used any strong systemic inducer of cytochrome P450 (CYP) 3A metabolism (e.g., rifampin, St John's wort) in the 3 months before visit 2.
* Patient has not complied with the requirements for restricted and prohibited medications and nonmedication therapies during the baseline period.

Recreational Drug Use:

* Patient has a positive drug screen for alcohol or recreational drugs (including cannabinoids) or nonprescribed controlled substances at screening (these assessments may be repeated once, after a reasonable time period at the investigator's discretion, but within the screening period) or at baseline.
* Patient has a history of alcohol or drug abuse/dependence/misuse within 1 year prior to screening.

General:

* Patient has any painful condition syndrome (e.g., neuropathy, fibromyalgia) or other concurrent medical or arthritic condition that has the potential to confound the assessment of pain in the index knee, in the investigator's opinion.
* Patient has a Hospital Anxiety and Depression Scale (HADS) score > 12 on either subscale at screening or baseline (visit 2 predose).
* Patient is involved in an ongoing or settled workers compensation claim, disability or litigation related to the index knee or any pain problem.
* Any condition that, in the investigator's opinion, makes the patient unsuitable for study participation.
* Patient is an employee of the Astellas Group, the Contract Research Organization (CRO) involved or the investigator site executing the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 4 in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Pain Subscale Score | Baseline and Week 4
  WOMAC is a tri-dimensional, self-administered, patient-centered health status questionnaire designed to capture the elements of pain, stiffness and physical function in participants with OA of the knee and/or hip joints. The questionnaire consists of 24 questions, which are divided into three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). Each question is scored using 11-point NRS scale ranging from 0 (none) to 10 (extreme). The pain subscale contains five questions that ask about pain during the last 48 hours caused by arthritis in the index knee. A negative change indicates a reduction/improvement from baseline.

SECONDARY OUTCOMES:
Change from Baseline to End of Treatment (EOT) in WOMAC Pain Subscale Score | Baseline and EOT (up to 4 weeks)
  WOMAC is a tri-dimensional, self-administered, patient-centered health status questionnaire designed to capture the elements of pain, stiffness and physical function in participants with OA of the knee and/or hip joints. The questionnaire consists of 24 questions, which are divided into three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). Each question is scored using 11-point Numerical Rating Scale (NRS) scale ranging from 0 (none) to 10 (extreme). The pain subscale contains five questions that ask about pain during the last 48 hours caused by arthritis in the index knee. A negative change indicates a reduction/improvement from baseline.
Change from Baseline to EOT in WOMAC Physical Function Subscale Score | Baseline and EOT (up to 4 weeks)
  WOMAC is a tri-dimensional, self-administered, patient-centered health status questionnaire designed to capture the elements of pain, stiffness and physical function in participants with OA of the knee and/or hip joints. The questionnaire consists of 24 questions, which are divided into three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). Each question is scored using 11-point NRS scale ranging from 0 (none) to 10 (extreme). The physical function subscale contains 17 questions that ask about the difficulty following daily physical activities. A negative change indicates a reduction/improvement from baseline.
Change from Baseline to EOT in WOMAC Stiffness Subscale Score | Baseline and EOT (up to 4 weeks)
  WOMAC is a tri-dimensional, self-administered, patient-centered health status questionnaire designed to capture the elements of pain, stiffness and physical function in participants with OA of the knee and/or hip joints. The questionnaire consists of 24 questions, which are divided into three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). Each question is scored using 11-point NRS scale ranging from 0 (none) to 10 (extreme). The stiffness subscale contains two questions that ask about stiffness during the last 48 hours caused by the arthritis. A negative change indicates a reduction/improvement from baseline.
Change from Baseline to EOT in WOMAC Total Score | Baseline and EOT (up to 4 weeks)
  WOMAC is a tri-dimensional, self-administered, patient-centered health status questionnaire designed to capture the elements of pain, stiffness and physical function in participants with OA of the knee and/or hip joints. The questionnaire consists of 24 questions, which are divided into three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). Each question is scored using 11-point NRS scale ranging from 0 (none) to 10 (extreme). The total score is the sum of scores from pain, physical function and stiffness subscales. Total score ranges from 0 to 30. A negative change indicates a reduction/improvement from baseline.
Change from Baseline to EOT in WOMAC Walking Pain Score | Baseline and EOT (up to 4 weeks)
  WOMAC is a tri-dimensional, self-administered, patient-centered health status questionnaire designed to capture the elements of pain, stiffness and physical function in participants with OA of the knee and/or hip joints. The questionnaire consists of 24 questions, which are divided into three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). Each question is scored using 11-point NRS scale ranging from 0 (none) to 10 (extreme). The walking pain score is based on question 1 of the questionnaire on pain when walking on a flat surface. A negative change indicates a reduction/improvement from baseline.
Change from Baseline to Weeks 1 and 2 in WOMAC Pain Subscale Score | Baseline and Weeks 1 and 2
  WOMAC is a tri-dimensional, self-administered, patient-centered health status questionnaire designed to capture the elements of pain, stiffness and physical function in participants with OA of the knee and/or hip joints. The questionnaire consists of 24 questions, which are divided into three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). Each question is scored using 11-point NRS scale ranging from 0 (none) to 10 (extreme). The pain subscale contains five questions that ask about pain during the last 48 hours caused by arthritis in the index knee. A negative change indicates a reduction/improvement from baseline.
Change from Baseline to Weeks 1, 2 and 4 in WOMAC Physical Function Subscale Score | Baseline and Weeks 1, 2, and 4
  WOMAC is a tri-dimensional, self-administered, patient-centered health status questionnaire designed to capture the elements of pain, stiffness and physical function in participants with OA of the knee and/or hip joints. The questionnaire consists of 24 questions, which are divided into three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). Each question is scored using 11-point NRS scale ranging from 0 (none) to 10 (extreme). The physical function subscale contains 17 questions that ask about the difficulty following daily physical activities. A negative change indicates a reduction/improvement from baseline.
Change from Baseline to Weeks 1, 2 and 4 in WOMAC Stiffness Subscale Score | Baseline and Weeks 1, 2, and 4
  WOMAC is a tri-dimensional, self-administered, patient-centered health status questionnaire designed to capture the elements of pain, stiffness and physical function in participants with OA of the knee and/or hip joints. The questionnaire consists of 24 questions, which are divided into three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). Each question is scored using 11-point NRS scale ranging from 0 (none) to 10 (extreme). The stiffness subscale contains two questions that ask about stiffness during the last 48 hours caused by the arthritis. A negative change indicates a reduction/improvement from baseline.
Change from Baseline to Weeks 1, 2 and 4 in WOMAC Total Score | Baseline and Weeks 1, 2, and 4
  WOMAC is a tri-dimensional, self-administered, patient-centered health status questionnaire designed to capture the elements of pain, stiffness and physical function in participants with OA of the knee and/or hip joints. The questionnaire consists of 24 questions, which are divided into three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). Each question is scored using 11-point NRS scale ranging from 0 (none) to 10 (extreme). The total score is the sum of scores from pain, physical function and stiffness subscales. Total score ranges from 0 to 30. A negative change indicates a reduction/improvement from baseline.
Change from Baseline to Weeks 1, 2 and 4 in WOMAC Walking Pain Score | Baseline and Weeks 1, 2, and 4
  WOMAC is a tri-dimensional, self-administered, patient-centered health status questionnaire designed to capture the elements of pain, stiffness and physical function in participants with OA of the knee and/or hip joints. The questionnaire consists of 24 questions, which are divided into three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). Each question is scored using 11-point NRS scale ranging from 0 (none) to 10 (extreme). The walking pain score is based on question 1 of the questionnaire on pain when walking on a flat surface. A negative change indicates a reduction/improvement from baseline.
Change from Baseline to Weeks 1, 2, 3, 4 and EOT in Mean Daily Average Pain Score Assessed by the Numerical Rating Scale | Baseline and Weeks 1, 2, 3, 4 and EOT (up to 4 weeks)
  The NRS is an 11-point scale used to capture the participant's average pain in the last 24 hours on a daily basis. This scale is composed of a single question and the score ranges from 0 to 10, where 0 anchors "no pain" and 10 anchors "pain as bad as you can imagine." The mean daily average NRS pain score was derived from the daily index knee pain ratings recorded by participants in an electronic diary (e-diary) on the last 4 days prior to randomization. A negative change indicates a reduction/improvement from baseline.
Change from Baseline Patient Global Assessment (PGA) at Weeks 1, 2, 4 and EOT | Baseline and Weeks 1, 2, 4 and EOT (up to 4 weeks)
  The PGA is an 11-point NRS scale used to capture the participant's overall impression at the time of the assessment in the index knee. This is a single question and the score ranges from 0 to 10, where 0 anchors "very good" and 10 anchors "very poor." A negative change indicates a reduction/improvement from baseline.
Percentage of Participants who Achieves ≥ 30% Decrease from Baseline to EOT in WOMAC Pain Subscale Score | Baseline and EOT (up to 4 weeks)
  This is the percentage of participants who has a reduction from baseline to EOT in WOMAC pain subscale score of ≥ 30%. WOMAC is a tri-dimensional, self-administered, patient-centered health status questionnaire designed to capture the elements of pain, stiffness and physical function in participants with OA of the knee and/or hip joints. The questionnaire consists of 24 questions, which are divided into three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). Each question is scored using 11-point NRS scale ranging from 0 (none) to 10 (extreme). The pain subscale contains five questions that ask about pain during the last 48 hours caused by arthritis in the index knee.
Percentage of Participants who Achieves ≥ 50% Decrease from Baseline to EOT in WOMAC Pain Subscale Score | Baseline and EOT (up to 4 weeks)
  This is the percentage of participants who has a reduction from baseline to EOT in WOMAC pain subscale score of ≥ 50%. WOMAC is a tri-dimensional, self-administered, patient-centered health status questionnaire designed to capture the elements of pain, stiffness and physical function in participants with OA of the knee and/or hip joints. The questionnaire consists of 24 questions, which are divided into three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). Each question is scored using 11-point NRS scale ranging from 0 (none) to 10 (extreme). The pain subscale contains five questions that ask about pain during the last 48 hours caused by arthritis in the index knee.
Number of Participants with Treatment-Emergent Adverse Events | From first dose of study drug up to 30 days after last dose of study drug (up to 8 weeks)
  A TEAE is defined as an adverse event (AE) which starts or worsens after the first dose of study drug until 30 days after taking the last dose of study drug. This includes abnormal laboratory tests, vital signs or electrocardiogram data that are defined as AEs if the abnormality induces clinical signs or symptoms, requires active intervention, interruption or discontinuation of study drug or is clinically significant in the investigator's opinion.
Number of Participants with an Affirmative Response in Columbia - Suicide Severity Rating Scale (C-SSRS): Suicidal Ideation | From first dose of study drug up to end of study (up to 8 weeks)
  C-SSRS is a questionnaire used for suicide assessment, where participants respond to these questions: (1) Wish to be dead; (2) Non-specific active suicidal thoughts; (3) Active suicidal ideation with any methods (not plan) without intent to act; (4) Active suicidal ideation with some intent to act, without specific plan; and (5) Active suicidal ideation with specific plan and intent.
Number of Participants with an Affirmative Response in CSSRS: Suicidal Behavior | From first dose of study drug up to end of study (up to 8 weeks)
  C-SSRS is a questionnaire used for suicide assessment, where participants respond to these questions: (1) Preparatory acts or behavior; (2) Aborted attempt; (3) Interrupted attempt; (4) Actual attempt; and (5) Completed suicide.
Number of Participants with an Affirmative Response in CSSRS: Suicidal Ideation or Behavior | From first dose of study drug up to end of study (up to 8 weeks)
  C-SSRS is a questionnaire used for suicide assessment, where participants respond to any one of the ten suicidal ideation and behavior questions.
Number of Participants with an Affirmative Response in CSSRS: Self-injurious Behavior without Suicidal Intent | From first dose of study drug up to end of study (up to 8 weeks)
  C-SSRS is a questionnaire used for suicide assessment, where participants respond to the question "Has subject engaged in Non-Suicidal Self-Injurious Behavior?"

CONTACTS AND LOCATIONS:
Overall Officials: Medical Officer, Study Director — Astellas Pharma Europe B.V.
Locations (34):
- Belgium (3):
  - Site BE32003, Leuven
  - Site BE32002, Merksem
  - Site BE32004, Yvoir
- Czechia (4):
  - Site CZ42006, Hradec Králové
  - Site CZ42003, Kunovice
  - Site CZ42002, Prague
  - Site CZ42005, Prague
- Germany (6):
  - Site DE49007, Bayern
  - Site DE49006, Berlin
  - Site DE49004, Deggingen
  - Site DE49003, Leipzig
  - Site DE49001, Magdeburg
  - Site DE49005, Munich
- Hungary (9):
  - Site HU36002, Baja
  - Site HU36008, Balatonfüred
  - Site HU36005, Békéscsaba
  - Site HU36007, Budapest
  - Site HU36006, Debrecen
  - Site HU36001, Esztergom
  - Site HU36003, Komárom
  - Site HU36009, Szeged
  - Site HU36004, Veszprém
- Spain (8):
  - Site ES34002, A Coruña
  - Site ES34001, Barakaldo
  - Site ES34008, Barcelona
  - Site ES34012, Barcelona
  - Site ES34003, Bilbao
  - Site ES34005, Madrid
  - Site ES34004, Santiago de Compostela
  - Site ES34010, Valencia
- United Kingdom (4):
  - Site GB44006, London
  - Site GB44011, North Shields
  - Site GB44010, Oxfordshire
  - Site GB44012, West Midlands

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Watt FE, Blauwet MB, Fakhoury A, Jacobs H, Smulders R, Lane NE. Tropomyosin-related kinase A (TrkA) inhibition for the treatment of painful knee osteoarthritis: results from a randomized controlled phase 2a trial. Osteoarthritis Cartilage. 2019 Nov;27(11):1590-1598. doi: 10.1016/j.joca.2019.05.029. Epub 2019 Jul 26. PMID 31356878
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=289